CLINICAL TRIAL: NCT07056946
Title: Supra Inguinal Fascia Iliaca Block Versus Ultrasound-guided Caudal Analgesia for Pediatrics Undergoing Anterior and Lateral Thigh Surgeries: A Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Suzan Adlan Abdelrahman, assistant professor, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AP2502-501-098-195
Record Dates: First submitted 2025-06-29; First posted 2025-07-09 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Cancer Bone
Keywords: Supra inguinal fascia iliaca Block ,Caudal Analgesia,Pediatrics
MeSH Terms: conditions — Bone Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group C: in this group children will receive US-guided caudal analgesia (CA) after GA. (Active Comparator): The caudal block will be performed by visualizing the sacral hiatus at the level of the sacral cornu after placing the probe transversely obtaining a short axis view
  Interventions: Other: Caudal Block Anesthesia
- Group B: in this group children will receive lower limb peripheral nerve blocks in the form of US (Experimental): With the patient in the proper position, the skin is disinfected and the transducer positioned to identify the femoral artery and the iliopsoas muscle and fascia iliaca. The transducer is moved laterally until the sartorius muscle is identified. After a skin wheal is made, the needle is inserted in-plane
  Interventions: Other: Fascia Iliaca Nerve Block

INTERVENTIONS:
Other: Fascia Iliaca Nerve Block — With the patient in the proper position, the skin is disinfected and the transducer positioned to identify the femoral artery and the iliopsoas muscle and fascia iliaca. The transducer is moved laterally until the sartorius muscle is identified. After a skin wheal is made, the needle is inserted in-plane
  Arms: Group B: in this group children will receive lower limb peripheral nerve blocks in the form of US
Other: Caudal Block Anesthesia — The caudal block will be performed by visualizing the sacral hiatus at the level of the sacral cornu after placing the probe transversely obtaining a short axis view, two hyperechoic lines will appear between the sacral cornu the superficial line is the sacrococcygeal ligament
  Arms: Group C: in this group children will receive US-guided caudal analgesia (CA) after GA.

SUMMARY:
patients will then be randomized in the two groups.

1. Group C: in this group children will receive US-guided caudal analgesia (CA) after GA. The caudal block will be performed
2. Group B: in this group children will receive lower limb peripheral nerve blocks in the form of US-guided fascia iliaca Block.

DETAILED DESCRIPTION:
After assessment of eligibility criteria, a clinical nurse independent of the protocol will obtain the randomization number and patients will then be randomized in the two groups. Treatment allocation will follow the order of a predetermined randomization list and will be generated using random blocks. Randomized will be done through computer program with patient blinded to the type of intervention (single blinded).

1. Group C: in this group children will receive US-guided caudal analgesia (CA) after GA. The caudal block will be performed by visualizing the sacral hiatus at the level of the sacral cornu after placing the probe transversely obtaining a short axis view, two hyperechoic lines will appear between the sacral cornu the superficial line is the sacrococcygeal ligament which will be pierced by the needle 22-gauge echogenic non-stimulating 5-cm needle (Ultraplex; B. Braun Medical Bethlehem PA, USA) using the out-of-plane approach. After confirming the absence of any blood or cerebrospinal fluid in the aspiration the caudal mixture (1 mL/kg of 0.25% bupivacaine a maximum volume of 20 mL will be used) will be injected.
2. Group B: in this group children will receive lower limb peripheral nerve blocks in the form of US-guided fascia iliaca Block.

American Society of Anesthiologists recommends monitors, intravenous line, and O2 (3 L/min) through the nasal cannula will be used. All blocks will be executed under the guidance of a 5-13 MHz linear ultrasound probe covered in a sterile sheath and attached to a Sonosite (M- Turbo; SonoSite Inc. Bothell WA USA) portable ultrasound machine. Preoperatively the maximum dose of bupivacaine will be calculated (2 mg/kg) so as not to exceed the dose during injection in either group.

ELIGIBILITY:
Inclusion Criteria:

* Age 1-12 years
* scheduled for anterior and lateral thigh Surgeries
* American Society of Anesthesiologists (ASA) physical status II or III

Exclusion Criteria:

* Refusal of parental consent
* Allergy to any local anesthetics

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 70 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
• Estimation of time of first rescue postoperative analgesia | 4 hours postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided